CLINICAL TRIAL: NCT03926884
Title: Evaluation of the Three-Seeds Mixture Treatment in Chronic Obstructive Pulmonary Disease Patients: A Pilot Study
Brief Title: Evaluation of the Three-Seeds Mixture Treatment in Chronic Obstructive Pulmonary Disease Patients
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Veterans Affairs Medical Center, Miami (U.S. Federal Agency)
Collaborators: Dr. Robert Jackson (Unknown)
Responsible Party: Principal Investigator, Fei Tang, Research Health Scientist, Veterans Affairs Medical Center, Miami
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: A1248
Record Dates: First submitted 2019-04-10; First posted 2019-04-25 (Actual); Last update posted 2019-04-25 (Actual); Status verified 2019-04

CONDITIONS: Cough
MeSH Terms: conditions — Cough

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Tea1 group (Experimental): This is the treatment group. This group will be taking 2 grams of the "three-seeds" mixture twice a day for three weeks.
  Interventions: Dietary Supplement: Three-seeds mixture
- Tea2 group (Placebo Comparator): This is the control group. This group will be taking 0.02 grams of the "three-seeds" mixture once a day for three weeks.
  Interventions: Dietary Supplement: Control

INTERVENTIONS:
Dietary Supplement: Three-seeds mixture — mixture of white mustard seeds, radish seeds and beefsteak plant (Korean perilla, a species of Perilla in the mint family, widely cultivated and edible for humans; a daily food for Korean people; many Japanese people drink as tea) seeds
  Arms: Tea1 group
Dietary Supplement: Control — warm water with negligible amount of the three-seeds mixture
  Arms: Tea2 group

SUMMARY:
The purpose of this study is to test whether the three-seeds mixture tea reduces sputum and/or cough in COPD patients, and if so, to evaluate whether the three-seeds mixture changes the lung microbiome.

ELIGIBILITY:
Inclusion Criteria:

1. Males or females ages 50-80 at the time of entry
2. Non-smoker for at least 1 year
3. Chronic bronchitis with Fev1 <80% and Fev1/ Fvc <0.7 and daily sputum production
4. Documentation of COPD. We define COPD as the presence of irreversible airflow obstruction, presence of emphysema on CT scan or both. This determination will be by the pulmonary physicians leading this study.
5. Ability and willingness to provide informed consent.

Exclusion Criteria:

1. Current Smoker 2. Asthma or other respiratory diseases 3. Frail patients (unintended weight loss, long term fatigue). 4. Patients with acute COPD exacerbation

-

Min Age: 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Estimated)
Dates: Start 2019-06-01 (Estimated); Primary Completion 2020-06-01 (Estimated); Study Completion 2020-06-30 (Estimated)

PRIMARY OUTCOMES:
Sputum and cough score | One month
  Sputum and cough measured by Cough and Sputum Assessment Questionnaire. The minimum score of this questionnaire is 0, and the maximum score is 100, with lower scores indicating higher symptom/impact levels. The total score will be reported. The score will be summed to a total score.

IPD SHARING:
Plan to Share IPD: No